CLINICAL TRIAL: NCT06499948
Title: A Unicentric, Randomized, Open-label, Cross-over Clinical Trial to Assess the Effect of Dapagliflozin, Spironolactone and Their Combination, When Added to Renin-Angiotensin System Blockade, on Lowering Urine Albumin-to-Creatinine Ratio in Adult Patients with Alport Syndrome
Brief Title: Albuminuria Lowering Effect of Dapagliflozin, Spironolactone and Their Combination in Adult Patients with Alport Syndrome (COMBINE-ALPORT)
Acronym: COMBINE-ALPORT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stefan Lujinschi (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Institutul Clinic Fundeni (Other)
Responsible Party: Sponsor-Investigator, Stefan Lujinschi, MD, PhD candidate, Institutul Clinic Fundeni
Organization: Institutul Clinic Fundeni (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 66035
Record Dates: First submitted 2024-07-07; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-05

CONDITIONS: Alport Syndrome; Thin Basement Membrane Disease; Alport Nephropathy
Keywords: Alport syndrome; Type IV collagen; Albuminuria; Chronic kidney disease; Monogenic kidney disorders; Glomerulopathy
MeSH Terms: conditions — Nephritis, Hereditary; Hematuria, Benign Familial; Albuminuria; Renal Insufficiency, Chronic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Timeline:
  * First visit - screening and eligibility: assessing eligibility and adjusting the renin-angiotensin-system inhibitor dose (2 weeks);
  * Second visit - stable dose of renin-angiotensin-system inhibitor (4 weeks);
  * Third visit - randomization: patients are randomized to receive either Spironolactone 25 mg od or Dapagliflozin 10 mg od (first treatment period: 4 weeks);
  * Fourth visit - first wash-out: the intervention is stopped (4 weeks);
  * Fifth visit - second treatment period: switching the treatment between the two groups (second treatment period: 4 weeks);
  * Sixth visit - second wash-out: the intervention is stopped (4 weeks);
  * Seventh visit - third treatment period: the whole cohort will receive the combined therapy consisting in Dapagliflozin 10 mg od and Spironolactone 25 mg od (4 weeks);
  * Eighth visit - third wash-out: the intervention is stopped (4 weeks);
  * Ninth visit - end of study: after the third wash-out period is finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Succession no.1: Spironolactone followed by Dapagliflozin followed by the combined therapy arm (Experimental): The patients will be randomized to receive either Spironolactone or Dapagliflozin on top of standard therapy (stable doses of renin-angiotensin-system inhibitors) in a crossover trial design (4 weeks of treatment followed by 4 weeks of wash-out). Finally, the whole cohort will receive both Spironolactone and Dapagliflozin for another 4 weeks.
  Treatment succession no.1 description: (1)1st treatment period - patients will receive Spironolactone 25 mg od on top of standard for 4 weeks; (2) 1st washout-period - treatment with Spironolactone will be stopped for 4 weeks; (3) 2nd treatment period - patients will receive Dapagliflozin 10 mg od for 4 weeks; (4) 2nd washout-period - treatment with Dapagliflozin will be stopped for 4 weeks; (5) 3rd treatment period - patients will receive Spironolactone 25 mg od plus Dapagliflozin 10 mg od for 4 weeks; (6) 3rd washout-period - treatment with Spironolactone and Dapagliflozin will be stopped for 4 weeks.
  Interventions: Drug: Treatment with Spironolactone followed by Dapagliflozin followed by their combination
- Succession no.2: Dapagliflozin followed by Spironolactone followed by the combined therapy arm (Experimental): The patients will be randomized to receive either Spironolactone or Dapagliflozin on top of standard therapy (stable doses of renin-angiotensin-system inhibitors) in a crossover trial design (4 weeks of treatment followed by 4 weeks of wash-out). Finally, the whole cohort will receive both Spironolactone and Dapagliflozin for another 4 weeks.
  Treatment succession no.2 description: (1) 1st treatment period - patients will receive Dapagliflozin 10 mg od on top of standard for 4 weeks; (2) 1st washout-period - treatment with Dapagliflozin will be stopped for 4 weeks; (3) 2nd treatment period - patients will receive Spironolactone 25 mg od for 4 weeks; (4) 2nd washout-period - treatment with Spironolactone will be stopped for 4 weeks; (5) 3rd treatment period - patients will receive Spironolactone 25 mg od plus Dapagliflozin 10 mg od for 4 weeks; (6) 3rd washout-period - treatment with Spironolactone and Dapagliflozin will be stopped for 4 weeks.
  Interventions: Drug: Treatment with Dapagliflozin followed by Spironolactone followed by their combination

INTERVENTIONS:
Drug: Treatment with Spironolactone followed by Dapagliflozin followed by their combination — After titrating the renin-angiotensin-system inhibitor dose, patients will receive 25 mg of Spironolactone once daily for 4 weeks. Spironolactone will be stopped after 4 weeks. The first treatment period will be followed by 4 weeks of wash-out. After the first wash-out period, treatment with Dapagliflozin will be started. Patients will receive 10 mg of Dapagliflozin once daily for 4 weeks. Dapagliflozin will be stopped after 4 weeks. The second treatment period will be followed by 4 weeks of wash-out. After the second wash-out period, treatment with both Spironolactone 25 mg and Dapagliflozin will be started. Patients will receive 25 mg of Spironolactone once daily in combination with 10 mg of Dapagliflozin daily for a duration of 4 weeks. Spironolactone and Dapagliflozin will be stopped after 4 weeks. The third treatment period will be followed by 4 weeks of wash-out, after which the study will be finalized.
  Other Names: Treatment succession no. 1; Spironolactone-Dapagliflozin-Combination; SDC succession; Spironolactone first
  Arms: Succession no.1: Spironolactone followed by Dapagliflozin followed by the combined therapy arm
Drug: Treatment with Dapagliflozin followed by Spironolactone followed by their combination — After titrating the renin-angiotensin-system inhibitor dose, patients will receive 10 mg of Dapagliflozin once daily for 4 weeks. Dapagliflozin will be stopped after 4 weeks. The first treatment period will be followed by 4 weeks of wash-out. After the first wash-out period, treatment with Spironolactone will be started. Patients will receive 25 mg of Spironolactone once daily for 4 weeks. Spironolactone will be stopped after 4 weeks. The second treatment period will be followed by 4 weeks of wash-out. After the second wash-out period, treatment with both Spironolactone and Dapagliflozin will be started. Patients will receive 25 mg of Spironolactone once daily in combination with 10 mg of Dapagliflozin daily for a duration of 4 weeks. Spironolactone and Dapagliflozin will be stopped after 4 weeks. The third treatment period will be followed by 4 weeks of wash-out, after which the study will be finalized.
  Other Names: Treatment succession no. 2; Dapagliflozin-Spironolactone-Combination; DSC succession; Dapagliflozin first
  Arms: Succession no.2: Dapagliflozin followed by Spironolactone followed by the combined therapy arm

SUMMARY:
Alport syndrome (AS) is one of the most common monogenic kidney disorders, oftentimes leading to end-stage kidney disease (ESKD). As AS is caused by variants involving type IV collagen genes (COL4), there is no specific treatment aimed at stopping the disease progression. Large studies have validated the use of renin-angiotensin-system inhibitors (RASis) in AS, as these drugs can slow the progression to chronic kidney disease (CKD). These studies included mainly pediatric patients with X-linked AS (XLAS). There is a lack of data regarding the therapeutic approach in patients having autosomal dominant AS (ADAS).

Recent data from murine studies suggest that the combined therapy using a sodium-glucose-cotransporter 2 inhibitor (SGLT2i) and a mineralocorticoid receptor blocker (MRB) can reduce proteinuria in COL4A3 knock-out mice. The albuminuria lowering effect of this combination was demonstrated in other non-diabetic nephropathies. Used in monotherapy, both drugs have showed protective and antifibrotic effects in murine models of AS.

The COMBINE-ALPORT trial aims to evaluate the albuminuria lowering effect of Dapagliflozin, Spironolactone and their combination in adult patients with genetically proven AS when added to maximum tolerated RASi dose. As proteinuria is the primary driver of CKD progression, and the change in albuminuria is widely used as a surrogate endpoint for kidney disease progression, lowering albuminuria will delay the onset of ESKD in patients with AS.

The main hypothesis of COMBINE-ALPORT trial is that the association of Dapagliflozin and Spironolactone will significantly reduce albuminuria in adult patient with AS.

The patients will be randomized to receive either Spironolactone or Dapagliflozin on top of standard therapy (maximum RASi dose) in a cross-over trial design (4 weeks of treatment followed by 4 weeks of wash-out). Finally, the whole cohort will receive both Spironolactone and Dapagliflozin for another 4 weeks.

The patients will visit the clinic every 4 weeks for checkups and tests.

The primary outcome is the effect on albuminuria by each treatment regimen (Spironolactone, Dapagliflozin or their combination).

ELIGIBILITY:
Inclusion Criteria:

* Genetically proven Alport syndrome (AS) - defined as following:

  * gt;Men having hemizygous pathogenic/likely pathogenic variants involving COL4A5 gene - classified as X-linked AS involving men
  * gt;Women having heterozygous pathogenic/likely pathogenic variants involving COL4A5 gene - classified as X-linked AS involving women
  * gt;Both men and women with heterozygous pathogenic/likely pathogenic variants involving COL4A3 or COL4A4 genes - classified as autosomal dominant AS
  * gt;Both men and women with homozygous pathogenic/likely pathogenic variants involving COL4A3 or COL4A4 genes - classified as autosomal recessive AS
  * gt;Patients having variants of uncertain significance will be included if the fulfill at least 2 of the following criteria: (1) clinical features suggestive of AS, (2) positive family history suggestive of AS (i.e., at least one grade I relative having the same variant and presenting clinical features suggestive of AS) and (3) kidney biopsy showing the characteristic lesion of AS (i.e., structural defect of the glomerular basement membrane, "basket-wave" appearance of the basement membrane, lamination of the basement membrane) or for thin basement membrane disease (i.e., diffusely thin basement membrane)
* Age between 18 and 70 years-old at the time of enrolment
* Baseline estimated glomerular filtration rate (eGFR) over 10ml/min/1.73m2 at the time of enrolment
* Stable kidney function: variation of eGFR under 25% from baseline in the last 6 weeks before randomization
* 24-hours urine albumin-to-creatinine ratio greater than 30 mg/g after adjusting the dose of renin-angiotensin-system inhibitor
* Stable renin-angiotensin-system inhibitor dose for at least 2 weeks before randomization

Exclusion Criteria:

* The need for kidney replacement therapy (i.e., hemodialysis, peritoneal dialysis, and kidney transplant) for more than 4 weeks in the last 12 months before enrollment
* Treatment with Spironolactone or Dapagliflozin for more than 14 days in the last 28 days prior to enrollment
* History of prior serious adverse event due to Spironolactone or Dapagliflozin
* Active neoplasia
* Autosomal dominant or recessive polycystic kidney disease
* Type I diabetes
* Patients with type II diabetes and diabetic nephropathy
* Diagnosis of another concomitant distinct glomerulopathy (with the exception of concomitant IgA nephropathy on kidney biopsy)
* Pregnancy and breastfeeding
* History of solid organ transplant
* Immunosuppressive treatment in the last 12 weeks prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hours urine albumin-to-creatinine ratio (UACR) compared to baseline after treatment with Dapagliflozin, Spironolactone and with their combination | 24-hours UACR will be measured at 0, 2, 6, 10, 14, 18, 22, 26 and 30 weeks after eligibility assessment

SECONDARY OUTCOMES:
Change in estimated glomerular filtration ratio (eGFR) compared to baseline after treatment with Dapagliflozin, Spironolactone and with their combination | eGFR will be measured at 0, 2, 6, 10, 14, 18, 22, 26 and 30 weeks after eligibility assessment
Change in serum potassium compared to baseline after treatment with Dapagliflozin, Spironolactone and with their combination | Serum K will be measured at 0, 2, 6, 10, 14, 18, 22, 26 and 30 weeks after eligibility assessment
The occurrence of adverse events, including serious adverse events | During and after each period of treatment, up to 24 weeks after randomization (30 weeks after assessing eligibility)
Change in urinary electrolytes excretion (sodium and potassium) compared to baseline after treatment with Dapagliflozin, Spironolactone and with their combination | Urinary sodium and potassium will me measured each 4 weeks up to 24 weeks after randomization: before and after each period of treatment and wash-out

OTHER OUTCOMES:
Reduction of 24-hours UACR with more than 30% from baseline after treatment with Dapagliflozin, Spironolactone and with their combination | Change of UACR will be asses after each period of treatment (at 4, 12 and 20 weeks after randomization)
Reduction of 24-hours UACR with more than 50% from after treatment with Dapagliflozin, Spironolactone and with their combination | Change of UACR will be asses after each period of treatment (at 4, 12 and 20 weeks after randomization)
Reduction of eGFR with more than 30% from baseline after treatment with Dapagliflozin, Spironolactone and with their combination | Change in eGFR will be asses after each period of treatment (at 4, 12 and 20 weeks after randomization)
Reduction of eGFR with more than 50% from baseline and/or doubling serum creatinine and/or initiation of kidney replacement therapy after treatment with Dapagliflozin, Spironolactone and with their combination | Change in eGFR will be asses after each period of treatment (at 4, 12 and 20 weeks after randomization)
Increase in serum potassium over 5.5 mmol/l and with more than 15% compared to baseline after treatment with Dapagliflozin, Spironolactone and with their combination | Changes in serum K will be assessed after each period of treatment (4, 12 and 20 weeks after randomization)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundeni Clinical Institute, Bucharest, Sector 2, Romania

IPD SHARING:
Plan to Share IPD: Undecided